CLINICAL TRIAL: NCT05359679
Title: Impact Collaboratory Transforming Dementia Care - Can Value Champions Reduce Inappropriate Prescribing for People With Dementia?
Brief Title: Can Value Champions Reduce Inappropriate Prescribing for People With Dementia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FY21_Demo2_Parchman; 5U54AG063546-03 (NIH)
Record Dates: First submitted 2022-03-14; First posted 2022-05-04 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Med: Dementia
Keywords: Prescribing
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a pragmatic cluster randomized trial across two Accountable Care Organizations. (ACOs) Within each ACO 15 primary care clinics will be randomized to the intervention arm or control arm of the study. From each intervention clinic, one clinician will participate in a clinical champion training program and subsequently work to decrease the prescribing of potentially inappropriate medications among patients with dementia among their colleagues. Medicare Part D pharmacy claims data will be analyzed at the end of the 12-month intervention for the primary outcome, the medication possession rates (MPR) for three groups of potentially inappropriate medications: antipsychotic medications, benzodiazepines, and hypoglycemic medications (sulfonylureas and insulin) among patients with a diagnosis of dementia.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Value Champion Training Program (Experimental): Intervention arm.
  Interventions: Behavioral: Value Champion Training Program
- Standard Care (Active Comparator): Control group.
  Interventions: Other: No Intervention

INTERVENTIONS:
Behavioral: Value Champion Training Program — Clinicians from primary care clinic sites randomized to the intervention arm of the study will complete a 6-month clinician value champion training program by participating in a series of 12 web-based training sessions. No intervention will be conducted at clinics in the control arm.
  Arms: Value Champion Training Program
Other: No Intervention — Usual clinical care - no value champion present at this clinical setting
  Arms: Standard Care

SUMMARY:
The primary objective is to assess the effectiveness of training a clinician to be a 'value champion' within clinical settings to decrease the use of three classes of potentially inappropriate prescription medications (PIMs) among people living with dementia (PLWD). Secondary objectives include determining if the intervention is associated with a reduction in emergency department (ED) visits or hospitalizations due to a fall, and examining five implementation outcomes: appropriateness, feasibility, fidelity, penetration, and equity.

This study is a pragmatic cluster-randomized trial to test the effectiveness of a primary care clinician value champion for de-implementing PIMs among patients 65 years of age and older with a diagnosis of dementia. Medicare Part D pharmacy claims data will be analyzed at the end of the 12-month intervention for the primary outcome, the medication possession rates (MPR) for three groups of potentially inappropriate medications: antipsychotic medications, benzodiazepines, and hypoglycemic medications (sulfonylureas and insulin). In a similar fashion, a hospital admission, or an emergency department visit for a fall will be assessed at the end of the intervention using Medicare claims data. Finally, the five implementation outcomes will be evaluated at the end of the intervention from notes entered by the value champions in project workbooks.

Primary care clinics within each of the two participating ACOs will be randomized to either the intervention or control arms of the study. Prior to random assignment, the investigators will stratify practices based on high versus low historic prescribing rates. A primary care clinician from each clinic selected for the trial in the intervention arm (n=30 across the two ACOs) will be recruited as a clinician value champion for each intervention clinic. The clinician value champion will participate in twice monthly value champion web-based training sessions for six months and then launch a 12-month initiative within the clinician value champions' clinics to reduce PIM prescribing among PLWD. Study outcomes will be assessed 12 months after the clinician value champions launch the initiative.

The hypothesis is that for each medication class, the intervention will produce clinically relevant decreases in mean possession rates of 10% of a standard deviation in patients seen in intervention clinics compared to those who are seen in control group clinics.

DETAILED DESCRIPTION:
Background on Condition, Disease, or Other Primary Study Focus:

For people living with dementia (PLWD) the overuse of Potentially Inappropriate Medications (PIMs), those for which the potential for harm outweighs benefit, remains a persistent problem despite evidence-based guidelines supporting de-adoption. A group of geriatric experts convened by the Choosing Wisely initiative identified three classes of PIMs for PLWD: antipsychotics, benzodiazepines, and hypoglycemics (sulfonylureas and insulin) with adequate glycemic control. In a systematic review the prevalence of PIMs when cognitive impairment was reported ranged from 20.6% to 80.5%. Approximately 14.3% of Medicare Part D enrollees with dementia residing in the general community are prescribed an antipsychotic. The prevalence of potentially inappropriate benzodiazepine prescriptions has been reported to be as high as 20% among elderly persons with dementia living in the community. The proportion of elderly patients with an A1c < 7% who received a prescription for sulfonylurea, insulin or combined insulin and sulfonylurea therapies was 35.2%, 24.2% and 16.3% respectively and was as prevalent in those with dementia as in those without. Park and colleagues compared rates of prescribing low-value medications in the elderly from 2006-2015 in both traditional Medicare and Medicare Advantage. Not only was there no difference in rates between the two groups, there was also no evidence of any decline in rates of prescribing over time, including use of benzodiazepines in PLWD.

Study Rationale:

The rationale for decreasing the use of PIMs is that use in this population of patients results in a greater likelihood of harm than benefit. Documented harms in the medical literature includes falls, worsening cognitive impairment, hospital admission, functional impairment, and death.

Name and Description of the Intervention:

One clinician value champion from each clinic randomized to the intervention arm will complete a value champion training program led by the P.I. and then implement care redesign activities in the clinical practice setting to reduce the use of low value prescribing in older adults with dementia. The 6-month training phase will consist of twice monthly web-based training sessions. A recently completed Robert Wood Johnson Foundation (RWJF)-funded Value Champion Fellowship program resulted in the development of a training curriculum comprised of 10 learning modules for the training phase of the intervention and a project workbook to guide clinician value champions during the 12-month project phase. Following the 6 months of training, clinician value champions will participate in a monthly 1-hour shared learning sessions via video conference to share successes, challenges, and brainstorm solutions for 12 months (months 10-22 of the study). The investigators will invite former value champion fellows and faculty from the RWJF fellowship to participate in these meetings to support this new cohort of value champions.

ELIGIBILITY:
Inclusion Criteria - clinician practices:

* Clinical practices with 3 or more primary care providers (defined as a primary care physician (specialty code of 08 or 11), nurse practitioner (specialty code = 50) or physician's assistant (specialty code = 97), and
* Clinical practices with clinical encounters with 10 or more Medicare beneficiaries with Alzheimer's or Alzheimer's related dementia in the base years (2019-2020).

Inclusion Criteria - Medicare beneficiaries:

* Seen by a clinician at a participating practice as evidenced by one or more evaluation and management claim,
* Continuous coverage in Medicare Parts A, B and D and no months of Part C (Medicare Advantage),
* Two or more claims with an International Statistical Classification of Diseases (ICD-10) diagnosis for Alzheimer's or Alzheimer's related dementia 30 days apart or 1 inpatient stay with a principal diagnosis of Alzheimer's.

Exclusion Criteria- Medicare beneficiaries:

* Medicare beneficiaries with a diagnosis of metastatic cancer or
* Medicare beneficiaries enrolled in hospice any time in the 6 months before the start of the intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorella Palazzo, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Tabata-Kelly M, Palazzo LG, Perloff J, Kiel L, Parchman M, Penfold RB. Champion-Led Deprescribing for Persons with Dementia in Primary Care: A Qualitative Study in Accountable Care Organizations. J Gen Intern Med. 2026 Feb 2. doi: 10.1007/s11606-026-10234-8. Online ahead of print. PMID 41629556
- [Derived] Parchman ML, Perloff J, Ritter G. Can clinician champions reduce potentially inappropriate medications in people living with dementia? Study protocol for a cluster randomized trial. Implement Sci. 2022 Sep 27;17(1):63. doi: 10.1186/s13012-022-01237-0. PMID 36163181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care clinics were randomized to intervention or control arms, stratified by high versus low historic prescribing rates of potentially inappropriate medications (PIMs).
  Patients accrued to the study according to the intervention arm clinic or control arm clinic where they were prescribed PIMs.
Pre-assignment Details: Value Champion clinicians (VCs) were enrolled and consented for the purpose of training activities, and for qualitative data collection only. No baseline or outcome data was collected for the VCs.
Units Other Than Participants: clinics
Groups:
- Value Champion: Intervention arm
  Primary care clinic sites were randomized to the intervention arm of the study. One clinician from each intervention site completed a 6-month clinician Value Champion training program by participating in a series of 12 web-based training sessions. Value Champions engaged with other clinicians at their site regarding deprescribing PIMs.
- Standard Care: Control arm
  No Intervention: Usual clinical care - no Value Champion present at this clinical setting
Period: Overall Study
Arm/Group | Value Champion | Standard Care
Started | 1613; 18 clinics | 1668; 17 clinics
Value Champion Clinicians | 19; 18 clinics | 0; 0 clinics
Completed | 1613; 18 clinics | 1668; 17 clinics
Not Completed | 0; 0 clinics | 0; 0 clinics

BASELINE CHARACTERISTICS:
Population: There were too few participants meeting inclusion criteria for analysis at one of the two study sites (site 2).
  1. Dementia prevalence was only 3% for site 2, vs 20% at site 1.
  2. By the time all exclusions and eligibility criteria were applied, the number of cases got even smaller;
  3. Site 2 data did not support reliable attribution to study national provider identification number (clinician identifier or NPI). We could not perform a meaningful analysis with site 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Value Champion Training Program | Standard Care | Total
Number analyzed (Participants) | 1570 | 1612 | 3182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1570 | 1612 | 3182
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1055 | 1182 | 2237
  Male | 515 | 430 | 945
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaskan Native | 0 | 0 | 0
  Asian/Pacific Islander | 21 | 51 | 72
  Black or African American | 305 | 372 | 677
  Hispanic | 37 | 46 | 83
  Non-Hispanic White | 1171 | 1091 | 2262
  Other/Unknown | 36 | 52 | 88

OUTCOME MEASURES:

1. Primary Outcome: Medication Possession Ratio (MPR) for Any Antipsychotics Medication
Description: The Medication Possession Ratio is calculated from Medicare Part D claims data as quotients with denominator equal to the length of the quarter and the numerators equal to the days supply for prescriptions within the medication class filled during the quarter, plus excess days-supply from the previous period minus excess days-supply remaining at the end.
Time Frame: 21 months
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Value Champion Training Program | Standard Care
Number analyzed (Participants) | 1570 | 1612
Medication possession ratio | 0.64 (0.079) | 0.56 (0.073)

2. Primary Outcome: Medication Possession Ratio (MPR) for Any Benzodiazepine Medication
Description: as for outcome 1
Time Frame: 21 months
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Value Champion Training Program | Standard Care
Number analyzed (Participants) | 1570 | 1612
Medication possession ratio | 0.29 (0.064) | 0.28 (0.074)

3. Primary Outcome: Medication Possession Ratio (MPR) for Insulin Medication
Description: as for outcome 1
Time Frame: 21 months
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Value Champion Training Program | Standard Care
Number analyzed (Participants) | 1570 | 1612
Medication possession ratio | 0.48 (0.094) | 0.43 (0.078)

4. Primary Outcome: Medication Possession Ratio (MPR) for Any Sulfonylureas Medications
Description: as for outcome 1
Time Frame: 21 months
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Value Champion Training Program | Standard Care
Number analyzed (Participants) | 1570 | 1612
Medication possession ratio | 0.51 (0.108) | 0.46 (0.065)

5. Secondary Outcome: Percent of Patients With Emergency Department (ED) Visits
Description: Mean percent of patients with Emergency Department (ED) visits in a given study follow up month
Time Frame: 21 months
Measure: Mean (Standard Deviation); unit: percentage of participants per month
Arm/Group | Value Champion Training Program | Standard Care
Number analyzed (Participants) | 1570 | 1612
percentage of participants per month | 8.1 (0.018) | 6.0 (0.016)

6. Secondary Outcome: Percentage of Falls
Description: Mean percentage of falls reported in claims in a given study month
Time Frame: 21 months
Measure: Mean (Standard Deviation); unit: percent of falls per month
Arm/Group | Value Champion Training Program | Standard Care
Number analyzed (Participants) | 1570 | 1612
percent of falls per month | 3.85 (1.5) | 4.47 (1.7)

ADVERSE EVENTS:
Time Frame: 10 months
Description: We surveyed clinical Value Champions administering the intervention monthly on whether any adverse events occurred with their patients receiving the intervention.
  All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not monitored/assessed in clinicians
Groups:
- Value Champion: Intervention arm:
  Primary care clinic sites were randomized to the intervention arm of the study. One clinician from each intervention site completed a 6-month clinician Value Champion training program by participating in a series of 12 web-based training sessions. Value Champions engaged with other clinicians at their site regarding deprescribing potentially inappropriate medications (PIMs).
Arm/Group | Value Champion | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/1613 | 0/1668
Serious Adverse Events (participants affected / at risk) | 0/1613 | 0/1668
Other Adverse Events (participants affected / at risk) | 2/1613 | 0/1668
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Value Champion (N=1613) | Standard Care (N=1668)
Worsening of diabetes control (Endocrine disorders) | 1 (1) | 0 (0)
Worsening of anxiety (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT05359679/Prot_SAP_000.pdf